CLINICAL TRIAL: NCT01287884
Title: Correlation of Arterial Blood Gas (ABG) and Venous Blood Gas (VBG) in the Undifferentiated Critically Ill Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 600824
Record Dates: First submitted 2011-01-31; First posted 2011-02-02 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-11

CONDITIONS: Patients Needing Blood Gases
Keywords: ABG; VBG; pH; pCO2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Venous Blood Gas (No Intervention): All subjects have an ABG and VBG drawn. No intervention.
  Interventions: Other: Venous Blood Gas

INTERVENTIONS:
Other: Venous Blood Gas — patients who have been identified by the treating physician as needing an ABG will receive an VBG is they consent to take part in the study

SUMMARY:
The primary objective of this study is to identify a correlation between the pH and pCO2 in arterial and venous blood. The secondary objectives include a correlation of pulse oximetry and arterial pO2 along with subgroup analyses of specific patient populations such as congestive heart failure, chronic obstructive pulmonary disease, diabetic ketoacidosis, pneumonia, overdose, and trauma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older Signed consent Patient in the ED or ICU Have a disease state that necessitates obtaining an ABG Have a disease state that necessitates pulse oximetry monitoring

Exclusion Criteria:

* Any contraindication to arterial or venous blood draw Prior enrollment in the study during the current hospitalization Pregnancy Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2010-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Degree to which pH and pCO2 correlate between ABG and VBG | 5 minutes
  ABG and VBG will be obtained 5 minutes apart and compared

CONTACTS AND LOCATIONS:
Overall Officials: Eli Zeserson, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Newark, Delaware, United States